CLINICAL TRIAL: NCT05509400
Title: BHV3000-406 (C4951004): A Phase 4, Randomized, Double-blind Placebo-Controlled, Efficacy and Tolerability Trial of Rimegepant for the Acute Treatment of Migraine in Adults Unsuitable for Triptan Use
Brief Title: Efficacy and Tolerability of Rimegepant for the Acute Treatment of Migraine in Adults Unsuitable for Triptan Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-406; C4951004 (Other: Alias Study Number); 2022-001175-14 (Registry Identifier: CTIS (EU)); 2024-513269-37-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: Migraine; Acute Migraine; Headache; Acute treatment of Migraine in adults unsuitable for triptans
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rimegepant (Experimental): Rimegepant - Double-blind (DB) Phase: One dose of rimegepant 75 mg Oral Disintegrating Tablet (ODT)
  Rimegepant/Rimegepant - Open-label Extension (OLE) Phase: participants receive one dose rimegepant 75 mg ODT as needed for a qualifying acute migraine. A qualifying migraine is an attack of moderate or severe headache pain intensity. Migraine headache pain intensity will be measured on a 4-point numeric rating scale (0=none, 1=mild, 2=moderate, 3=severe)
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): Placebo - Double-blind (DB) Phase: One dose of matching placebo
  Placebo/Rimegepant - Open-label Extension (OLE) Phase: participants receive one dose rimegepant 75 mg ODT for a qualifying migraine
  Interventions: Drug: Placebo; Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — DB Phase: Rimegepant 75 mg Orally Disintegrating Tablet (ODT)
  Arms: Rimegepant
Drug: Placebo — DB Phase: matching placebo
  Arms: Placebo
Drug: Rimegepant — OLE Phase: Rimegepant 75 mg ODT in association with each of the first 5 qualifying migraines

SUMMARY:
This study is being conducted to evaluate the efficacy and tolerability of rimegepant in a population of adults that are unsuitable for triptan medications due to a previous intolerance, lack of efficacy, or contraindication (including a history of clinically-relevant cardiovascular disease).

DETAILED DESCRIPTION:
This study is being conducted to evaluate the efficacy and tolerability of rimegepant in a population of adults that are unsuitable for triptan medications due to a previous intolerance, lack of efficacy, or contraindication (including a history of clinically-relevant cardiovascular disease). Rimegepant will be further evaluated in this population with as needed use in a 12-week, open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age.
* Migraine attacks, on average, lasting about 4 - 72 hours if untreated.
* 4 to 14 migraine days per month on average across the 3 months prior to the Screening Visit (month is defined as 28 days for the purpose of this protocol).
* Less than 15 headache days (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and throughout the Screening Phase.
* Subjects must be able to distinguish migraine attacks from tension/cluster headaches.
* Subjects on prophylactic migraine medication (excluding CGRP antagonists) are permitted to remain on therapy if they have been on a stable dose for at least 3 months (12 weeks) prior to the Screening Visit, and if the dose is not expected to change during the course of the study.
* Triptan unsuitable

Exclusion Criteria:

-Target Disease Exclusion:

1. History of cluster headache, basilar migraine, or hemiplegic migraine
2. Current medication overuse headaches
3. Headaches occurring 15 or more days per month (migraine or non-migraine) in any of the 3 months prior to the Screening Visit
4. Active chronic pain syndrome (such as fibromyalgia, chronic pelvic pain, complex regional pain syndrome [CRPS])
5. Other pain syndromes (including trigeminal neuralgia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, interfere with study assessments of safety or efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of rimegepant with placebo in the acute treatment of migraine, as measured by migraine headache pain relief at 2-hours post-dose during the Double-Blind Treatment (DBT) Phase. | 2 hours post-dose
  Migraine headache pain relief will be assessed using the percentage of subjects with a headache pain intensity of none or mild. Migraine headache pain intensity will be measured on a 4-point numeric rating scale (0=none, 1=mild, 2=moderate, 3=severe).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- United States (23):
  - Clinical Research Institute, Los Angeles, California
  - Ki Health Partners LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Wr-Msra, Llc, Lake City, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites Network - Ormond Clinical Research Unit, Ormond Beach, Florida
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Collective Medical Research, Overland Park, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Community Clinical Research Network Inc, Marlborough, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Rochester Medical Group, Rochester Hills, Michigan
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Clinvest Research, LLC, Springfield, Missouri
  - St Charles Clinical Research, Weldon Spring, Missouri
  - DM Clinical Research - NY, NY, Brooklyn, New York
  - New York Neurology Associates, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
  - Red Star Research, LLC, Lake Jackson, Texas
  - DM Clinical Research, Tomball, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (2):
  - USC Clinical Trials Centre, Sippy Downs, Queensland
  - Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Medical University Innsbruck, Innsbruck, Tyrol
- Belgium (5):
  - Cabinet Privé Dr. Simona Sava, Saint-Nicolas, Liège
  - GZA Ziekenhuizen, Antwerp
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
- Canada (5):
  - University of Calgary South Health Campus, Calgary, Alberta
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Clinique Neuro-Lévis, Lévis, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - ALPHA Recherche Clinique, Québec
- Denmark (3):
  - University Hospital of Southern Denmark, Esbjerg
  - Danish Headache Center, Glostrup Municipality
  - Hospitalsenhed Midt, Viborg
- Finland (4):
  - Helsinki Headache Center, Helsinki, Uusimaa
  - Terveystalo Ruoholahti, Helsinki
  - Terveystalo Tampere Rautatienkatu, Tampere
  - Terveystalo Pulssi, Turku
- France (8):
  - Timone Hospital, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hospices Civils de Lyon - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Annecy Genevois, Epagny Metz-Tessy
  - CHU de Lille - Hôpital Salengro, Lille
  - CHU Nice Hopital Cimiez, Nice
  - Hopital Lariboisiere, Paris
  - CHU Saint-Etienne - Hopital Nord, Saint-Etienne
- Germany (4):
  - Neurologische Praxis Prof. Dr. Hartmut Gobel, Kiel, Schleswig-Holstein
  - University Hospital Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Neurologische Ambulanz, Kopfschmerzambulanz, Berlin
  - Kopfschmerzzentrum Frankfurt, Frankfurt
- Italy (7):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - AOU Luigi Vanvitelli, Napoli, Naples
  - Fondazione Policlinico Campus BioMedico, Rome, RM
  - Foundation IRCCS Neurological Institute Carlo Besta, Milan
  - AOU Policlinico di Modena, Modena
  - Fondazione Mondino - Istituto Neurologico Nazionale IRCCS, Pavia
  - Headache and Pain Unit - IRCCS San Raffaele, Rome
- Mexico (4):
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Centro de Investigación Médica de Aguascalientes (CIMA), Aguascalientes
  - Operadora Unidad de Investigación En Salud de Chihuahua, Sa de Cv, Mexico City
  - Clinstile SA de CV, Mexico City
- Poland (11):
  - Centrum Medyczne Neuromed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól, Lubusz Voivodeship
  - Concept Medica, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Damiana Walbrzyska, Warsaw, Masovian Voivodeship
  - Instytut Zdrowia dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim, Małopolska
  - Vita Longa Sp. Z o.o., Katowice
  - MICS Centrum Medyczne Szczecin, Szczecin
  - Praktyka Lekarska, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Centrum Leczenia Bolu dr n med Lukasz Kmieciak, Lodz, Łódź Voivodeship
- Spain (5):
  - University Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Virgen del Rocio University Hospital, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- Sweden (5):
  - CTC Solna, Solna, Stockholms LÄN [se-01]
  - CTC Uppsala, Uppsala, Uppsala County
  - Skåneuro Privatmottagning, Lund
  - Hälsoklustret, Stockholm
  - Akardo MedSite, Stockholm
- United Kingdom (5):
  - Re: Cognition Health Ltd., Edgebaston, Birmingham
  - 4 Medical Clinical Solutions London, Ilford, Essex
  - Lakeside Healthcare Group Research, Corby, Northamptonshire
  - Kings College London, London
  - 4 Medical Clinical Solutions, Swinton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ashina M, McAllister P, Gaul C, Leyva-Rendon A, Ramirez LM, Nalpas C, Thiry A, Abraham L, Fountaine RJ, Fullerton T. Rimegepant for acute treatment of migraine in triptan-unsuitable adults: A randomized, double-blind, placebo-controlled phase 4 trial. Cephalalgia. 2025 Nov;45(11):3331024251395298. doi: 10.1177/03331024251395298. Epub 2025 Nov 18. PMID 41255093
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-406